CLINICAL TRIAL: NCT01725035
Title: The Role of Hepatic De Novo Lipogenesis (DNL) in the Pathogenesis of Hepatic Steatosis in Obese Children and Adolescents
Brief Title: Hepatic De Novo Lipogenesis (DNL)in the Pathogenesis of Hepatic Steatosis in Obese Youth
Acronym: DNL
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: American Heart Association (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1008007192; 11CRP5620013 (Other Grant/Funding Number: American Heart Association); 1R01DK114504-01A1 (NIH)
Record Dates: First submitted 2012-10-30; First posted 2012-11-12 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Hepatic Steatosis; Fatty Liver
Keywords: De Novo Lipogenesis; Fatty Liver; Hepatic Steatosis; Gene variants
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fatty liver
- Non Fatty liver

SUMMARY:
Nonalcoholic Fatty Liver Disease (NAFLD) is becoming the most common cause of liver disease in pediatrics, but little is known about its pathophysiology in children. While studies in obese adults with hepatic steatosis have described an increased hepatic de novo lipogenesis (DNL) depending on the diet, there are no studies exploring the mechanisms by which excess hepatic triglycerides increases in obese youths, thus explaining the accompanying dyslipidemia and the metabolic syndrome. The central hypothesis of this study is that hepatic conversion of carbohydrates to lipid (DNL) is enhanced and associated with accumulation of excess liver fat, dyslipidemia and hepatic insulin resistance in obese youths with hepatic steatosis. The overall goal is to examine whether hepatic DNL is increased in obese youths with steatosis compared to matched controls without steatosis.

Hypotheses: Hepatic conversion of carbohydrates to lipid (DNL) is enhanced and is associated with accumulation of excess liver fat, dyslipidemia and hepatic insulin resistance in obese youths with hepatic steatosis.

DETAILED DESCRIPTION:
In this study obese youths, adolescents and young adults (12-30 years) will undergo MRI (magnetic resonance imaging) measurement of liver lipid content to determine hepatic fat content. They will undergo a sugary drink (75 grams of glucose and 25 grams of fructose) challenge and Hepatic de novo lipogenesis will be determined as the incorporation of deuterium, from deuterium labeled water (D2O), into plasma triglycerides. Subjects will undergo a 6 hours study assessing de novo lipogenesis, an oral glucose tolerance test, dual energy x-ray absorptiometry, magnetic resonance imaging, and Euglycemic-Hyperinsulinemic Clamp.

This study record has been re-opened in 2019 and updated to reflect any changes having remained open since its inception with the Yale University IRB and also having obtained additional funding though NIDDK.

ELIGIBILITY:
Inclusion Criteria:

* Cases will meet the following criteria:

  * BMI higher than 75th percentile
  * Hepatic fat fraction (the amount of fat into the liver) greater or equal than 5.5%
  * Absence of any endocrinopathy
  * Absence of any therapy with medication known to alter glucose metabolism

Controls will meet the following criteria:

* BMI higher than 75th percentile
* Hepatic fat fraction (the amount of fat into the liver) lower than 5.5%
* Absence of any endocrinopathy
* Absence of any therapy with medication known to alter glucose metabolism
* Absence of any therapy with medication known to alter glucose metabolism

Exclusion Criteria:

* BMI under the 75th percentile
* Hepatic fat fraction (the amount of fat into the liver) less than 5.5%
* Absence of any endocrinopathy
* Any therapy with medication known to alter glucose metabolism

Controls will meet the following criteria:

* BMI under the 75th percentile
* Hepatic fat fraction (the amount of fat into the liver) greater than or equal to 5.5%
* Any endocrinopathy
* Any therapy with medication known to alter glucose metabolism

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The majority of the research subjects will be recruited from the Yale Pediatric Obesity Clinic and the Endocrine Clinic. Following the oral glucose tolerance test (OGTT):normal glucose tolerant if plasma glucose at two hours is <140 mg/dl and impaired glucose tolerant if plasma glucose is ≥140 mg/dl. All subjects must be in good general health, have a normal medical history and physical exam, and have no endocrinopathies or other diseases that might affect glucose metabolism. They will not be on any medications that are known to alter glucose or insulin metabolism or certain psychiatric medications. Subjects determined to be eligible will receive a MRI to determine Hepatic Fat Content. Subjects will agree to genetic testing to determine genotype.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
de novo lipogenesis response to high carbohydrate meal in obese kids with fatty liver | Study visit 3

SECONDARY OUTCOMES:
de novo lipogenesis response to high carbohydrate meal in obese kids without fatty liver | Study visit 3

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Caprio, M.D., Principal Investigator — Yale University; Nicola Santoro, M.D./Ph.D,, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States